CLINICAL TRIAL: NCT06866119
Title: Effects of Estrogen Replacement on Cardiometabolic Endpoints in Women With Primary Ovarian Insufficiency
Brief Title: Effects of Estrogen on Heart Health in Women With Primary Ovarian Insufficiency
Acronym: ENCODE
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara L. Stockman, MD, PhD, Endocrine Fellow, Massachusetts General Hospital
Other Study IDs: 2025P000601; GR1000466 (Other Grant/Funding Number: Massachusetts General Hospital - Division of Endocrinology)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Primary Ovarian Insufficiency; Premature Menopause; Metabolic Complications; Endothelial Function (FMD); Estrogen Replacement Therapy
Keywords: primary ovarian insufficiency; premature menopause; estrogen replacement therapy; cardiovascular disease prevention; POI; ERT
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case participants with Primary Ovarian Insufficiency: This group is comprised of women (assigned female at birth), age 30-40yo who have a clinically documented diagnosis of primary ovarian insufficiency (POI) within 6 months and be planning to clinically initiate estrogen replacement therapy (with 100mcg transdermal 17beta-estradiol twice weekly and micro-ionized progesterone either 100mg daily or 200mg cyclically) with their own provider. Women in the group may not be on systemic estrogen, progesterone or testosterone therapy, have contraindications for estrogen administration or known atherosclerotic cardiovascular disease or equivalents. They must also not take lipid lowering therapy or antihypertensive or anti-inflammatory/immune suppressant medications or be pregnant or breastfeeding. After a telephone screen to determine eligibility, the group will engage in two in-person study visits. The first occurs prior to the initiating estrogen replacement therapy and the second after 6 months of treatment.
- Health control participants without Primary Ovarian Insufficiency: This group is compromised of women (assigned female at birth), age 30-40yo who have regular menstrual cycles every 21-35 days. Women in the group may not be on systemic estrogen, progesterone or testosterone therapy, have contraindications for estrogen administration or known atherosclerotic cardiovascular disease or equivalents. They must also not take lipid lowering therapy or antihypertensive or anti-inflammatory/immune suppressant medications or be pregnant or breastfeeding. After a telephone screen to determine eligibility, the group will in a single in-person study visit.

SUMMARY:
The goal of this observational study is to study the effects of treating women with Primary Ovarian Insufficiency (POI) with estrogen replacement therapy to bolster the evidence backing cardiometabolic preventive care in women with POI. The main question it aims to answer is:

Does 6 months of estrogen replacement therapy for women with POI improved markers of heart health?

Women newly diagnosed with POI (within 6 months) who are planning to start estrogen replacement therapy from their clinical provider will undergo assessment of markers of heart health before and after 6 months of treatment. These markers will also be compared to those obtained from healthy women without POI.

DETAILED DESCRIPTION:
Primary Ovarian Insufficiency (POI) is known to adversely affect bone and CV health. Despite the established role for ERT in bone health and the potential cardioprotection suggested by recent studies, few women with POI receive treatment. In this proposed study, we aim to characterize potential salient short-term benefits of ERT on CV surrogates. We hypothesize that among women newly diagnosed with POI, clinical initiation of ERT with transdermal estrogen will improve cardiometabolic risk surrogates, including endothelial function. This study will enhance the body of evidence underpinning guideline-directed approaches to cardiometabolic preventive health care for women with POI.

For this observational study, women newly diagnosed with POI (within 6 months) who are planning to clinically initiate hormonal replacement with 100mcg transdermal 17beta-estradiol twice weekly and micro-ionized progesterone (either 200mg cyclically or 100mg daily) will undergo assessment of cardiometabolic endpoints before and after 6 months of treatment. For comparison, healthy women without POI matched 1:1 on age, BMI, and PREVENT™ risk score category (low-high risk) will undergo parallel assessments at baseline.

Participants will undergo a medical history, physical exam, anthropomorphic measurements, blood sampling, brachial artery flow-mediated dilation (FMD), as a measure of peripheral endothelial function relevant to development of incident CVD, and whole-body DXA to assess body composition. Case participants with POI will participate in two in-person study visits that occur just prior to initiation of ERT and 6-months into treatment. Healthy control participants only participate in a single baseline visit.

The primary endpoint will be brachial artery flow-mediated dilation (FMD). Secondary endpoints will include measures of metabolic dysregulation (possibly including, but not limited to, hemoglobin A1c, circulating lipid levels, HOMA-IR for insulin resistance and DEXA-derived visceral adipose tissue) and characterization of circulating immune/inflammatory biomarkers (possibly including, but not limited to, CRP and pro-inflammatory cytokines IL-6 and TNF-α).

ELIGIBILITY:
Inclusion criteria (I):

* female sex
* age 30-40
* CASE PARTICIPANTS ONLY: clinically documented POI diagnosis within 6 months
* CASE PARTICIPANTS ONLY: planning to clinically initiate 100mcg transdermal 17beta-estradiol twice weekly and micro-ionized progesterone (either 100mg daily or 200mg cyclically)
* CONTROL PARTICIPANTS ONLY: regular menstrual cycles every 21-35 days

Exclusion criteria (E):

* CASE PARTICIPANTS ONLY: genetic POI etiology
* CASE PARTICIPANTS ONLY: any prior initiation of ERT
* systemic estrogen, progesterone or testosterone therapy within the past 6 months (including contraception, except for locally acting intrauterine devices - IUDs)
* lipid lowering therapy within the past 6 months
* use of antihypertensive medication within the past 6 months
* current treatment with prescription, systemic (oral, IV, or IM) steroids or anti-inflammatory/immune suppressant medical therapies (excluding topical therapies, UV therapy, ASA-derivative therapies, or NSAIDS) for autoimmune/inflammatory diseases (psoriasis, RA, IBD, lupus), post-transplant care, asthma, or pain syndromes
* use of oral steroids or prescription oral anti-inflammatory/immune suppressant medication for >7 days within the past 1 month
* use of IV or IM steroids or IV or IM anti-inflammatory/immune suppressant medication within the past 3 months
* self-reported history of breast and/or estrogen dependent malignancy
* self-reported history of deep vein thromboembolism, pulmonary embolism or stroke
* self-reported severe liver disease such as cirrhosis
* self-reported hypercoagulable disorder
* uncontrolled hypertension at baseline Visit #1- systolic blood pressure (SBP) ≥180 and/or diastolic blood pressure (DBP) ≥110
* tobacco use within 6 months
* self-reported history of myocardial infarction, stroke, coronary revascularization or diabetes as a CVD risk equivalent
* stable or unstable angina
* self-reported history of heart failure
* pregnancy or breastfeeding
* concurrent enrollment in conflicting research study

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals assigned female at birth are eligible to participate in the study regardless of gender. However, participants may not be on systemic estrogen, progesterone or testosterone therapy, aside from the relevant prescribed estrogen replacement therapy for those with POI.
Study Population: The study population is comprised of women newly diagnosed with POI (within 6 months) who are planning to clinically initiate hormonal replacement with 100mcg transdermal 17beta-estradiol twice weekly and micro-ionized progesterone (either 200mg cyclically or 100mg daily). For comparison, healthy women without POI matched 1:1 on age, BMI, and PREVENT™ risk score category (low-high risk) will also be studied.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Brachial artery Flow Mediated Vasodilation (FMD) | 6 months
  Brachial artery flow-mediated dilation (FMD) is a non-invasive measure of endothelial function relevant to the development of incident cardiovascular disease. Brachial artery FMD will be reported as a percentage (%FMD), calculated by comparing the change in brachial artery diameter during reactive hyperemia to the baseline diameter. %FMD will be compared between case participants with POI and healthy control participants at baseline. The change in %FMD after 6 months of estrogen replacement therapy will be determined for case participants with POI.

SECONDARY OUTCOMES:
Metabolic biomarkers | 6 months
  Urine and serum biomarkers relating to metabolism (including glucose and lipid metabolism, body composition)
Immune/inflammatory biomarkers | 6 months
  Urine and serum biomarkers relating to inflammation and immune activation

CONTACTS AND LOCATIONS:
Overall Officials: Markella V. Zanni, MD, Study Chair — MGH/HMS
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Plans are for IPD to be shared to the NIH BioLINCC data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available 12 months after study completion and will remain available for a duration of time consonant with NIH policies.
Access Criteria: Access criteria are as per the NIH BioLINCC data repository.